CLINICAL TRIAL: NCT04230252
Title: A Single-dose, Open-label, Randomized, Two-treatment, Two-period, Crossover Study in Healthy Subjects to Assess the Bioequivalence of the Newly Formulated Tylenol® Tablet (Acetaminophen) to the Tylenol® 8H ER Tablet (Acetaminophen) Under Fasting Conditions
Brief Title: A Study of the Newly Formulated Tylenol Tablet (Acetaminophen) to the Tylenol 8 Hour (H) Extended Release (ER) Tablet (Acetaminophen) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR108737; RWJ3465PAI1001 (Other: Janssen Korea, Ltd., Korea); DDS19-028BE (Other: Janssen Korea Ltd. Korea)
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence 1: Reference Drug + Test Drug (RT) (Experimental): Participants will receive 8 hour (H) extended-release (ER) acetaminophen tablet orally in period 1 (Reference) followed by newly formulated acetaminophen tablet orally in period 2 (Test). Each period will be separated by a washout period of at least 7 days.
  Interventions: Drug: Acetaminophen
- Treatment Sequence 2: Test Drug + Reference Drug (TR) (Experimental): Participants will receive newly formulated acetaminophen tablet orally in period 1 (Test) followed by 8 hour ER acetaminophen tablet orally in period 2 (Reference). Each period will be separated by a washout period of at least 7 days.
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen — Acetaminophen tablet will be administered orally in treatment sequence 1 and 2.
  Other Names: Tylenol; JNJ-28678-AAA

SUMMARY:
The purpose of this study is to evaluate the bioequivalence of the newly formulated Tylenol tablet (acetaminophen 650 mg) with respect to the Tylenol 8 Hour (H) Extended Release (ER) tablet (acetaminophen 650 mg) in healthy participants under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening. If there are abnormalities, they must be consistent with the underlying illness in the study population. This determination must be recorded in the participant's source documents
* Healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel including liver enzymes, other specific tests, hematology, urinalysis or breathing alcohol test are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* Blood pressure (after the participant is sitting for 5 minutes) between 90 and 140 millimeters of Mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic
* Have no history of psychiatric disorder within the 5 years prior to the screening
* Have no history of gastrointestinal resection that may affect drug absorption

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency (creatinine clearance below 60 milliliter per minute [mL/min]), thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Clinically significant abnormal physical examination, vital signs, or 12 lead ECG at screening as deemed appropriate by the investigator
* Known allergies, hypersensitivity, or intolerance to acetaminophen or its excipients
* History of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which is considered cured with minimal risk of recurrence)
* Taken any disallowed therapies as noted in local prescribing information, concomitant therapy before the planned first dose of study drug

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Analyte Concentration (Cmax) | Up to 24 hours post-dose
  Cmax is the maximum observed analyte concentration.
Area Under the Concentration-time Curve From Time 0 to Time of the Last Measurable Concentration (AUC [0-last]) | Up to 24 hours post-dose
  AUC (0-last) is the area under the concentration-time curve from time 0 to time of the last measurable concentration (non-below quantitation limit).

SECONDARY OUTCOMES:
Area Under the Concentration-time Curve From Time 0 to Infinite Time (AUC[0-infinity]) | Up to 24 hours post-dose
  AUC(0-infinity) is the area under the concentration-time curve from time 0 to infinite time, calculated as the sum of AUC (0-last) and C(last)/lambda(z).
Percentage of Area Under the Concentration-time Curve Extrapolated from Last Measurable Concentration to Infinite Time (Extrapolated %AUCinfinity) | Up to 24 hours post-dose
  Percentage of area under the concentration-time curve extrapolated from last measurable concentration to infinite time (extrapolated %AUCinfinity) is calculated using formula: (AUC [0-infinity] minus AUC [0-last]/AUC [0-infinity])*100.
Time to Reach the Maximum Observed Analyte Concentration (Tmax) | Up to 24 hours post-dose
  Tmax is the time to reach the maximum observed analyte concentration.
Time to Last Measurable Plasma Concentration (T [last]) | Up to 24 hours post-dose
  Tlast is the time to last measurable plasma concentration.
Elimination Rate Constant (Lambda [z]) | Up to 24 hours post-dose
  Lambda (z) is the apparent terminal elimination rate constant determined by linear regression using the terminal log-linear phase of the log transformed concentration-time curve.
Elimination Half-Life (t 1/2) | Up to 24 hours post-dose
  t1/2 is defined as apparent is associated terminal elimination half-life associated with the terminal slope (lambda [z]) of the semilogarithmic drug concentration-time curve, calculated as: 0.693/lambda(z).
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 41 days
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea
Locations (1):
- H plus Yangji Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency